CLINICAL TRIAL: NCT05295862
Title: Giessen Acute Stroke Registry
Brief Title: Giessen Stroke Registry
Acronym: GIST
Status: Recruiting | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Tobias Braun, Senior Physician, University of Giessen
Other Study IDs: GI-NEU-2101
Record Dates: First submitted 2022-02-14; First posted 2022-03-25 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Stroke, Acute; Comorbidities and Coexisting Conditions; Critical Care
Keywords: Acute Stroke; Comorbidities; Clinical Management
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the planned study project is to assess the current situation regarding the treatment of patients with stroke. Specifically, various treatment strategies are to be associated and correlated with clinical endpoints, mortality or functional outcome in order to generate arguments for or against individual aspects of therapy. The focus will be on unresolved treatment approaches in acute therapy (e.g. periprocedural management, such as blood pressure, blood glucose, temperature, or airway management, during recanalizing therapies) as well as in secondary prevention on the stroke unit or intensive care unit, such as starting point, mode, and dosage of antithrombotic therapies.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death worldwide as well as the most common cause of permanent disability (Baron 1999).

In the acute phase of ischemic cerebral infarction, the goal of therapy is the rapid reopening of the occluded vessel. This should restore blood flow to the inferiorly supplied brain tissue surrounding the infarct core, the penumbra, and limit the extent of the irreversibly damaged infarct core (Astrup 1981). According to the current guidelines for acute therapy of ischemic stroke, thrombolysis with recombinant tissue-type plasminogen activator (rt-PA) can be performed within the first 4.5 hours after symptom onset (Ringleb 2015). The safety and efficacy of this therapy is considered proven (Hacke 2008, Wahlgren 2008). Outside this "time window", the incidence of bleeding complications increases.

In recent years, the efficacy of interventional reopening of an occluded vessel in combination with rt-PA or without rt-PA has additionally been demonstrated. Since the publication of the results of the landmark studies on thrombectomy (MR-CLEAN [Berkhemer 2014] ESCAPE [Goyal 2015], EXTEND-IA [Campbell 2015], SWIFT-PRIME [Saver 2015], REVASCAT [Jovin 2015]) in 2016 and a meta-analysis of these studies (Goyal 2016), this therapy is widely used in specialized centers. This intervention is also available outside the 4.5-hour time window when specialized imaging is used to visualize potentially salvageable brain tissue and thus patient selection. This can be done using perfusion imaging in computed tomography (CT) or magnetic resonance imaging (MRI). Here, a difference ("mismatch") between cerebral regional blood flow (CBF) and cerebral regional blood volume (CBV) represents potentially salvageable tissue (CBV/CBF mismatch). Similarly, structural brain imaging with MRI cannot yet detect irreversibly damaged tissue, as diffusion-weighted sequences show ischemia shortly after symptom onset, but fluid attenuated inversion recovery (FLAIR) sequences show ischemia after 4-6 hours (DWI-FLAIR mismatch). Also, salvageable tissue can be assumed in the presence of largely unremarkable imaging and high disease severity (clinical-imaging mismatch). Considering the risk of bleeding in larger already demarcated infarcts, systemic intravenous thrombolysis can also be added if necessary. In all mismatch situations, superiority of thrombolysis and thrombectomy has recently been demonstrated (Barow 2019).

The cornerstone of stroke therapy is the stroke unit concept. Diagnostics, acute therapy, secondary prophylaxis, and early rehabilitation treatment are coordinated in a specialized stroke unit. Depending on the hospital structure, acute diagnosis and therapy may also take place in an emergency room facility. The stroke unit concept is based on structured, interdisciplinary collaboration between neurologists, neuroradiologists, internists, neurosurgeons, speech therapists, occupational and physical therapists, nursing staff and the emergency medical services. Treatment in such a stroke unit alone reduces mortality by 18-46 percent relatively (3 percent absolutely), the risk of functional dependence by 29 percent, and the need for nursing home care or total home care by 25 percent (Stroke Unit Trialists Collaboration 2007). Key mechanisms of action appear to include careful adjustment of vital signs. Deviations in body temperature, blood glucose, and blood pressure lead to worse clinical outcomes (Sandercock 2008, Langhorne 2002, Sobesky 2009). In addition, patients should be screened early for dysphagia, i.e., swallowing disorders, and nutrition should be adjusted, which is a mandatory measure on stroke units (Sobesky 2009).

The background of the planned project is that although there has been an enormous increase in knowledge in the treatment of stroke patients in recent years based on prospective randomized trials (especially the establishment of thrombectomy in the acute phase as well as pioneering therapies in secondary prevention, e.g., treatment of patients with atrial fibrillation or persistent foramen ovale), many questions in the everyday practical implementation of these study results remain unresolved.

The aim of this research project is to generate new evidence for or against common treatment algorithms in fields where no randomized data are available. Among other things, it will be analyzed to what extent different preclinical algorithms (e.g., drip-and-ship management (i.e., secondary transfer of acutely ill patients from external hospitals to a center for thrombectomy), intraclinical treatment pathways, and early management on stroke units and intensive care units affect outcomerelevant parameters. The overall aim is to improve the current level of evidence on the management of stroke patients by analyzing a large database of individualized patient data.

The aim of the present - noninterventional and purely descriptive - project is to record treatment parameters of consecutive patients with stroke and to correlate them with clinical end points.

Specifically, a retrospective evaluation of patients who were hospitalized at the Department of Neurology due to stroke between the years 2018 and 2020 will be performed first. Specifically, it is planned to first identify these patients through a controlling query. Subsequently, various clinical parameters from the routine acute phase will be collected by reviewing the in-house electronic data systems. Aspects of data protection will be observed according to the local institutional guidelines. In order to analyze the outcome of the patients, contact will be made by means of a written questionnaire sent by mail, and subsequently, if necessary, by a telephone call. By providing the enclosed patient information and patient consent, the patient or legal guardian gives consent (or refusal) to the partial aspect of the telephone interview for the purpose of recording long-term outcome. . Patients who are deceased or cannot be reached will be included in the database without recording long-term outcome. Here, no clarification is provided.

In a second step, emerging aspects and treatment approaches resulting from the exploratory data analysis will also be recorded prospectively in the sense of a continuous expansion of the registry. If new approaches arise for the routine care of patients, such as adjustment of treatment algorithms, these can be evaluated first. Depending on the question, it may also be necessary to extend the period for retrospective evaluation of routine data in order to obtain a sufficient number of cases; in this case, the ethics committee will be informed.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Patient admitted for acute stroke (Stroke Unit or Intensive Care Unit)
* Informed Consent

Exclusion Criteria:

* Inclusion criteria not met

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted for acute stroke
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin-scale after 3 months | 3 months after initial stroke
  Funtional Outcome measured by modified Rankin-scale.
  The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Modified Rankin-scale after 12 months | 12 months after initial stroke
  Funtional Outcome measured by modified Rankin-scale.
  The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

SECONDARY OUTCOMES:
Intrahospital Mortality | Up to 6 weeks after initial stroke.
  Number of patients that died during initial hospital phase.
Short-term and long-term mortality | 3 months and 12 after initial stroke
  Number of patients that died over the course of 3 and 12 months
New stroke | 3 and 12 months after initial Stroke
  Number of patients with new stroke.

OTHER OUTCOMES:
Recurring pneumonia during follow-up | 3 and 12 months after initial Stroke
  Number of patients with recurring pneumonia.
Epilepsy | 3 and 12 months after initial Stroke
  Number of patients with occurence of epilepsy and its treatment
Cognitive decline | 3 and 12 months after initial Stroke
  Number of patients with cognitive decline as measured with the Montreal Cognitive Assessment
Tracheostomy | 3 and 12 months after initial Stroke
  Number of patients with need for longterm tracheostomy
Non-oral feeding | 3 and 12 months after initial Stroke
  Number of patients with need for longterm non-oral feeding
Reduction of quality of life | 3 and 12 months after initial Stroke
  Rate of reduction in quality of life as measured by the EQ-5D.
  High values represent a marked reduction in the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Braun, M.D., Principal Investigator — University of Giessen
Locations (1):
- Universitätsklinikum Gießen, Giessen, Hesse, Germany

REFERENCES:
- [Background] Baron JC. Mapping the ischaemic penumbra with PET: implications for acute stroke treatment. Cerebrovasc Dis. 1999 Jul-Aug;9(4):193-201. doi: 10.1159/000015955. PMID 10393405
- [Background] Astrup J, Siesjo BK, Symon L. Thresholds in cerebral ischemia - the ischemic penumbra. Stroke. 1981 Nov-Dec;12(6):723-5. doi: 10.1161/01.str.12.6.723. No abstract available. PMID 6272455
- [Background] Ringleb P., Köhrmann M., Jansen O., et al.: Akuttherapie des ischämischen Schlaganfalls, S2e-Leitlinie, 2021, in:Deutsche Gesellschaft für Neurologie (Hrsg.), Guidelines for Diagnostics und Therapy in Neurology.
- [Background] Hacke W, Kaste M, Bluhmki E, Brozman M, Davalos A, Guidetti D, Larrue V, Lees KR, Medeghri Z, Machnig T, Schneider D, von Kummer R, Wahlgren N, Toni D; ECASS Investigators. Thrombolysis with alteplase 3 to 4.5 hours after acute ischemic stroke. N Engl J Med. 2008 Sep 25;359(13):1317-29. doi: 10.1056/NEJMoa0804656. PMID 18815396
- [Background] Wahlgren N, Ahmed N, Davalos A, Hacke W, Millan M, Muir K, Roine RO, Toni D, Lees KR; SITS investigators. Thrombolysis with alteplase 3-4.5 h after acute ischaemic stroke (SITS-ISTR): an observational study. Lancet. 2008 Oct 11;372(9646):1303-9. doi: 10.1016/S0140-6736(08)61339-2. Epub 2008 Sep 12. PMID 18790527
- [Background] Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama a Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 2015 Jan 1;372(1):11-20. doi: 10.1056/NEJMoa1411587. Epub 2014 Dec 17. PMID 25517348
- [Background] Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 2015 Mar 12;372(11):1009-18. doi: 10.1056/NEJMoa1414792. Epub 2015 Feb 11. PMID 25671797
- [Background] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Background] Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GW, Cognard C, Cohen DJ, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Baxter BW, Devlin TG, Lopes DK, Reddy VK, du Mesnil de Rochemont R, Singer OC, Jahan R; SWIFT PRIME Investigators. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. N Engl J Med. 2015 Jun 11;372(24):2285-95. doi: 10.1056/NEJMoa1415061. Epub 2015 Apr 17. PMID 25882376
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Stroke Unit Trialists' Collaboration. Organised inpatient (stroke unit) care for stroke. Cochrane Database Syst Rev. 2013 Sep 11;2013(9):CD000197. doi: 10.1002/14651858.CD000197.pub3. PMID 24026639
- [Background] Sandercock PA, Counsell C, Gubitz GJ, Tseng MC. Antiplatelet therapy for acute ischaemic stroke. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD000029. doi: 10.1002/14651858.CD000029.pub2. PMID 18646056
- [Background] Langhorne P, Pollock A; Stroke Unit Trialists' Collaboration. What are the components of effective stroke unit care? Age Ageing. 2002 Sep;31(5):365-71. doi: 10.1093/ageing/31.5.365. PMID 12242199
- [Background] Ahmed N, Wahlgren N, Brainin M, Castillo J, Ford GA, Kaste M, Lees KR, Toni D; SITS Investigators. Relationship of blood pressure, antihypertensive therapy, and outcome in ischemic stroke treated with intravenous thrombolysis: retrospective analysis from Safe Implementation of Thrombolysis in Stroke-International Stroke Thrombolysis Register (SITS-ISTR). Stroke. 2009 Jul;40(7):2442-9. doi: 10.1161/STROKEAHA.109.548602. Epub 2009 May 21. PMID 19461022
- [Background] Barow E, Thomalla G. [Acute treatment of ischemic stroke : Current standards]. Nervenarzt. 2019 Oct;90(10):979-986. doi: 10.1007/s00115-019-0776-5. German. PMID 31407046
- [Background] Sobesky J. [Therapy of acute ischemic stroke]. Internist (Berl). 2009 Nov;50(11):1218-26. doi: 10.1007/s00108-009-2470-3. German. PMID 19838656